CLINICAL TRIAL: NCT00002413
Title: An Open Label Study of MKC-442 in at Least Triple Drug Combination in Patients Previously Treated With Nucleoside Reverse Transcriptase and Protease Inhibitors and Who Are Naive to Non-Nucleoside Reverse Transcriptase Inhibitors
Brief Title: A Study of MKC-442 in HIV-Positive Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Triangle Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 292B; MKC-304
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-04

CONDITIONS: HIV Infections
Keywords: Anti-HIV Agents; Viral Load; MKC 442
MeSH Terms: conditions — HIV Infections | interventions — emivirine

INTERVENTIONS:
Drug: Emivirine

SUMMARY:
The purpose of this study is to see if it is safe and effective to give MKC-442 plus at least two other anti-HIV drugs to patients who have never been treated with nonnucleoside reverse transcriptase inhibitors but who have been treated with nucleoside reverse transcriptase inhibitors and protease inhibitors. This study also determines how long a drug combination including MKC-442 is effective.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

Based on medical history, medical condition, prior use of antiretroviral drugs, and genotypic analysis of the predominant strain of HIV-1 isolated from plasma, administration of at least 2 available antiviral agents by prescription may be given with MKC-422.

Patients must have:

- HIV infection with HIV-1 RNA greater than or equal to 2,000 by Roche Amplicor method, within 30 days of entry.

Prior Medication:

Allowed:

* Prior nucleoside reverse transcriptase and protease inhibitors.
* Cytotoxic chemotherapy more than 30 days prior to entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Malabsorption or severe chronic diarrhea within 30 days prior to entry, or inability to consume adequate oral intake because of chronic nausea, emesis, or abdominal or esophageal discomfort.
* Inadequately controlled seizure disorder.
* Acute and clinically significant medical event within 30 days of screening.
* Any clinical or laboratory abnormality greater than Grade 3 toxicity, with the exception of the listed laboratory values.

Prior Medication:

Excluded:

* Non-nucleoside reverse transcriptase inhibitor therapy.
* Any unapproved experimental antiretroviral therapy.

Prior Treatment:

Excluded:

* Radiation therapy within 30 days of entry, except to a local lesion.
* Transfusion of blood or blood products within 21 days of screening.

Risk Behavior:

Excluded:

Active substance abuse that may interfere with compliance or protocol evaluations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult